CLINICAL TRIAL: NCT06688019
Title: A Comparison of High-flow Nasal Oxygen and Conventional Nasal Cannula in Monitored Anesthesia Care for Endoscopic Submucosal Dissection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2024-1108
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Patients Undergoing Endoscopic Submucosal Dissection
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Intervention Model Description: Arm 1: conventional nasal cannula group Arm 2: high-flow humidified oxygen-delivery system (OptiFlow THRIVE) group
Masking Description: Patients will be randomly allocated to 2 groups using computer-generated randomization method. Neither participants nor physicians will be blinded to the groups because of organizational reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional oxygenation (nasal cannula) arm (Experimental): conventional oxygenation arm will receive oxygen at 2L/min via nasal cannula
  Interventions: Device: conventional oxygenation (nasal cannula)
- high-flow humidified oxygen-delivery system (OptiFlow THRIVE) arm (Experimental): Optiflow THRIVE arm will receive oxygen at 50 L/min via Optiflow THRIVE
  Interventions: Device: high-flow humidified oxygen-delivery system (OptiFlow THRIVE)

INTERVENTIONS:
Device: conventional oxygenation (nasal cannula) — conventional oxygenation arm will receive oxygen at 2 L/min via nasal cannula, while Optiflow THRIVE arm will receive oxygen at 50 L/min via Optiflow THRIVE during the procedure.
  Arms: conventional oxygenation (nasal cannula) arm
Device: high-flow humidified oxygen-delivery system (OptiFlow THRIVE) — conventional oxygenation arm will receive oxygen at 2 L/min via nasal cannula, while Optiflow THRIVE arm will receive oxygen at 50 L/min via Optiflow THRIVE during the procedure.
  Arms: high-flow humidified oxygen-delivery system (OptiFlow THRIVE) arm

SUMMARY:
Sedation for endoscopic submucosal dissection places patients at risk of desaturation, and high-flow nasal oxygen may reduce the risk. The aim of this study is to evaluate the role of high-flow nasal oxygen during endoscopic submucosal dissection. We will compare the incidence of hypoxemia (defined as SpO2 lower than 90%) of conventional nasal oxygen cannula group and that of high-flow humidified oxygen-delivery system group during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo endoscopic sumucosal dissection under remimazolam-based sedation

Exclusion Criteria:

* dementia or cognitive dysfunction
* altered mental status
* intubated patients or tracheostomy
* pregnancy
* recent history of nasal bleeding
* contraindication for positive pressure ventilation
* patients under oxygen therapy
* illiteracy or foreigner

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-10-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxemia (SpO2 lower than 90%) measured with pulse oximetry during the procedure | during the procedure (from the start to the end of the endoscopic submucosal dissection), 1hour
  We will record the incidence of hypoxemia during the procedure.

SECONDARY OUTCOMES:
the number and duration of hypoxemia | during the procedure (from the start to the end of the endoscopic retrograde cholangiopancreatography), 1hour
  We will compare the number and duration of hypoxemia, the lowest SpO2 during procedure, need for airway intervention, the end tidal CO2 at the end of the procedure between the two groups.
the lowest SpO2 during procedure | during the procedure (from the start to the end of the endoscopic retrograde cholangiopancreatography), 1hour
  We will compare the number and duration of hypoxemia, the lowest SpO2 during procedure, need for airway intervention, the end tidal CO2 at the end of the procedure between the two groups.
need for airway intervention | during the procedure (from the start to the end of the endoscopic retrograde cholangiopancreatography), 1hour
  We will compare the number and duration of hypoxemia, the lowest SpO2 during procedure, need for airway intervention, the end tidal CO2 at the end of the procedure between the two groups.
the end tidal CO2 at the end of the procedure | during the procedure (from the start to the end of the endoscopic retrograde cholangiopancreatography), 1hour
  We will compare the number and duration of hypoxemia, the lowest SpO2 during procedure, need for airway intervention, the end tidal CO2 at the end of the procedure between the two groups.

IPD SHARING:
Plan to Share IPD: Undecided